CLINICAL TRIAL: NCT00293891
Title: A Study to Assess the Safety and Effectiveness of Tacrolimus Cream in the Treatment of Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: Astellas Pharma US, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 04-0-206
Record Dates: First submitted 2006-02-16; First posted 2006-02-20 (Estimated); Last update posted 2007-12-24 (Estimated); Status verified 2007-12

CONDITIONS: Psoriasis
Keywords: Treatment Outcome; Tacrolimus; Safety; Psoriasis
MeSH Terms: conditions — Psoriasis

INTERVENTIONS:
Drug: Tacrolimus Cream

SUMMARY:
A study to assess the safety and effectiveness of tacrolimus cream in the treatment of psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of plaque psoriasis

Exclusion Criteria:

* Skin disorder other than plaque psoriasis in the areas to be treated.
* Disease on only elbows, knees, and scalp

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 658 (Actual)
Dates: Study Completion 2007-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: J. Rico, MD, Study Director — Astellas Pharma US, Inc.
Locations (33):
- United States (27):
  - Birmingham, Alabama
  - Little Rock, Arkansas
  - San Diego, California
  - Denver, Colorado
  - Miami, Florida
  - West Palm Beach, Florida
  - Newnan, Georgia
  - Indianapolis, Indiana
  - Louisville, Kentucky
  - North Andover, Massachusetts
  - Ann Arbor, Michigan
  - Port Huron, Michigan
  - St Louis, Missouri
  - Omaha, Nebraska
  - New York, New York
  - Durham, North Carolina
  - Columbus, Ohio
  - Dayton, Ohio
  - Portland, Oregon
  - Knoxville, Tennessee
  - Dallas, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah
  - Norfolk, Virginia
  - Seattle, Washington
  - Milwaukee, Wisconsin
- Canada (6):
  - Calgary, Alberta
  - Edmonton, Alberta
  - Surrey, British Columbia
  - Moncton, New Brunswick
  - Laval, Quebec
  - Montreal, Quebec